CLINICAL TRIAL: NCT00449891
Title: Neuropsychological and Neuroanatomical Studies of Young Children With and Without Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: William E And Aenid R Weisgerber Foundation (Other)
Responsible Party: Principal Investigator, Tandy Aye, Assistant Professor, Stanford University
Other Study IDs: IRB 97517; 1102002-100-GHATW
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is being conducted to see if Type 1 diabetes mellitus has any affect on learning, behavior and development in young children and whether there are associated changes on their MRI scan.

DETAILED DESCRIPTION:
In this pilot study approximately 10-20 children between the ages of 3 to 10 years with Type 1 diabetes mellitus will have neuropsychological testing and a nonsedated MRI scan of the head performed every three years for three years. We will compare this to a control group of 10 children between the ages of 3 adn 10 years without Type 1 diabetes mellitus. The control subjects will neuropsychological testing and a nonsedated MRI scan of the head once. The children with Type 1 diabetes mellitus will not have any changes made to their current diabetes regimen.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for study subjects:

* To be between ages 3 to 10 years
* Have been diagnosed with type 1 diabetes for at least 6 months; and
* Do not have plans to move out of the area within the next 36 months.

Inclusion Criteria for control subjects:

* To be between ages 3 to 10 years

Exclusion Criteria:

* No history of head trauma with any loss of consciousness,
* Cystic fibrosis,
* Prematurity (born less than 30 weeks of gestation),
* Significant developmental delay (lack of single word speech or ability to walk independently by 18 months of age),
* Neurologic disease independent of diabetes (eg seizure disorder); or
* Medical contraindication to MRI procedure (eg metal appliances such as braces).

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: please see inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tandy Aye, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Aye T, Barnea-Goraly N, Ambler C, Hoang S, Schleifer K, Park Y, Drobny J, Wilson DM, Reiss AL, Buckingham BA. White matter structural differences in young children with type 1 diabetes: a diffusion tensor imaging study. Diabetes Care. 2012 Nov;35(11):2167-73. doi: 10.2337/dc12-0017. Epub 2012 Sep 10. PMID 22966090
- See also: Stanford University Division of Pediatric Endocrinology website — http://dped.stanford.edu